CLINICAL TRIAL: NCT04446949
Title: Documenting the Undocumented - The Use of Maternal Health Care and Pregnancy Outcomes in Undocumented Migrant Women in Norway.
Brief Title: Maternal Health Care and Pregnancy Outcomes in Undocumented Migrant Women in Norway.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Women's Public Health Association (NKS) (Unknown); Oslo Church City Mission (Unknown); Red Cross (Unknown); Department of Emergency General Practice (DEGP) Oslo and Bergen (Unknown)
Responsible Party: Principal Investigator, Cecilie Dahl, Dr. Cecilie Dahl, University of Oslo
Other Study IDs: 68329
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Transients and Migrants; Primary Health Care; Pregnancy Outcome
Keywords: Norway; Emergency care; Medical Birth Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Undocumented migrants
  Interventions: Other: Register follow-up
- Immigrants with Norwegian ID
  Interventions: Other: Register follow-up
- Norwegian residents
  Interventions: Other: Register follow-up

INTERVENTIONS:
Other: Register follow-up — Number of adverse pregnancy outcomes

SUMMARY:
Little research on the health service utilization and the health situation of undocumented pregnant migrants has been performed previously, and it is essential to obtain more information on the services given, and to examine whether residency status is a risk factor in maternal and perinatal health among migrants.This project will give new knowledge on undocumented women seeking care at the voluntary clinics and the emergency clinics (DEGPs) in Oslo and Bergen, their health care needs, and the medical follow-up they are provided. The project will present new knowledge by showing trends in undocumented pregnant migrants care seeking compared to general trends among other migrants and Norwegian residents. It will also give new knowledge on pregnancy outcomes and perinatal health in undocumented migrants compared to foreign and Norwegian born women. This approach has not previously been used to study undocumented migrants in Norway, and there are very few similar studies in other European countries. Cause and effect relations are rarely claimed in findings from observational epidemiologic studies, however the information from three different sources (voluntary clinics, emergency clinics and Medical Birth Registry) will give an overall picture of the use of primary health care in undocumented pregnant migrants, as well as a comparative assessment of maternal outcomes in this population. The proposed research will also give important knowledge on how to conduct quantitative research in a population that is difficult to reach, and that is not commonly included in research.

DETAILED DESCRIPTION:
Research questions and objectives

1. Work package 1 (WP1): What characterizes pregnant undocumented migrants attending the voluntary clinics in Oslo and Bergen from 2009 to 2020?

   1. Give a descriptive summary of the population of pregnant undocumented migrants seeking care (e.g. age, number of children, time stayed in Norway, work status, family network) and the medical problems they are presenting.
   2. Investigate the care received based on indicators such as number of antenatal visits and the extent of collaboration with or referral to other health facilities.
   3. Investigate the risk of pregnancy related complications (e.g. pre-eclampsia and gestational diabetes) and adverse perinatal outcomes (e.g. use of Caesarean Section and pre-term birth) in women seeking care at the clinics.
2. Work package 2 (WP2): Are there any consultation trends in pregnant undocumented migrants seeking emergency care at the emergency units (DEGPs) in Oslo and Bergen from 2007 to 2020?

   1. Give a descriptive summary of the population of undocumented migrants seeking emergency care at the DEGPs, in particular pregnant undocumented migrants seeking care.
   2. Investigate trends in emergency consultations at the DEGPs for pregnant undocumented migrants after the start of the voluntary clinics (2009/2014), comparing with the trends in consultations for the general population of pregnant women seeking care.
   3. Investigate trends in emergency consultations at the DEGPs for pregnant undocumented migrants after the start of the voluntary clinics (2009/2014), comparing to the trends in consultations for other undocumented migrants.
3. Work package 3 (WP3): What is the occurrence of pregnancy-related complications and adverse perinatal outcomes (as reported in the Medical Birth Registry of Norway) in patients without national identity number from 1999 to 2020?

   1. Investigate the prevalence of pregnancy related complications (e.g. pre-eclampsia, gestational diabetes, nutrient deficiency) in undocumented migrant women compared to foreign and Norwegian born women.
   2. Investigate the incidence of adverse perinatal outcomes (e.g. use of Caesarean section, pre-term birth, small for gestational age, low Apgar score) in undocumented migrant women compared with foreign and Norwegian born women.

ELIGIBILITY:
Inclusion Criteria:

* No registered Norwegian identity number
* Female

Exclusion Criteria:

* Male

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women giving birth in Norway
Study Population: WP1: Women attending voluntary clinics for primary care to undocumented migrants in Oslo and Bergen WP2: Patients without a national ID receiving treatment at the emergency care units in Oslo and Bergen WP3: Women registered to give birth in the Medical Birth Registry of Norway (probably undocumented migrants without a Norwegian ID, Norwegian residents with an immigration background, Norwegian-born women)
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adverse pregnancy outcomes | 1999-2020
  From medical records and the Medical Birth Registry
Primary health care use by undocumented pregnant migrants | 2007-2020
  From voluntary clinics and emergency units

SECONDARY OUTCOMES:
Health care use of undocumented migrants in general | 2007-2020
  From voluntary clinics and emergency units

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Dahl, PhD, MPH, Principal Investigator — University of Oslo

IPD SHARING:
Plan to Share IPD: No
We are not allowed to share IPD due to GDPR regulations and Norwegian Law.